CLINICAL TRIAL: NCT00118417
Title: Treatment Refractory Panic Disorder
Brief Title: Therapies for Treatment-Resistant Panic Disorder Symptoms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Naomi M. Simon, Director, Center for Anxiety and Traumatic Stress Disorders, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K23MH001831 (NIH); K23MH001831 (NIH); DSIR AT-CD
Record Dates: First submitted 2005-07-06; First posted 2005-07-11 (Estimated); Results first posted 2009-07-28 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Panic Disorder
Keywords: Selective serotonin reuptake inhibitor; Anxiety; Pharmacotherapy; Cognitive behavioral therapy; CBT
MeSH Terms: conditions — Panic Disorder; Anxiety Disorders | interventions — Clonazepam; Sertraline; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Participants in phase II will receive sertraline, or an equivalent medication, up to 100 mg plus a placebo pill. Participants in phase III will receive the same medication with cognitive behavioral therapy.
  Interventions: Drug: Sertraline; Behavioral: Cognitive behavioral therapy
- 2 (Experimental): Participants in phase II will receive sertraline, or equivalent medication, up to 200 mg. Participants in phase III they will receive the same medication with flexible clonazepam augmentation.
  Interventions: Drug: Clonazepam; Drug: Sertraline

INTERVENTIONS:
Drug: Clonazepam — Participants will receive clonazepam.
  Arms: 2
Drug: Sertraline — Participants will receive sertraline.
Behavioral: Cognitive behavioral therapy — Participants will receive cognitive behavioral therapy
  Arms: 1

SUMMARY:
This study will determine the effectiveness of different treatments for panic disorder symptoms in individuals who still have symptoms after initial treatment with medication.

DETAILED DESCRIPTION:
Panic disorder is a serious condition that may cause significant psychological and physical distress. Many patients with panic disorder remain symptomatic despite initial intervention. Unfortunately, little data is available to guide health care providers in "next-step" treatment approaches. This study will evaluate the effectiveness of treatments for individuals with panic disorder that is resistant to initial treatment with selective serotonin reuptake inhibitors (SSRIs).

This study will last 24 weeks and will comprise three phases. In Phase 1, participants will receive the SSRI sertraline for 6 weeks. Phase 1 will be used to determine participants' resistance to treatment. During Phase 1, participants will begin a medication schedule and symptom diary and will have weekly study visits to assess regimen adherence and any side effects they may be experiencing. In Phase 2, participants will be randomly assigned to 6 weeks of one of two treatments: sertraline at an elevated dose from that given in Phase 1 or a sertraline and placebo regimen. During Phase 2, participants will have 3 study visits. Self-report scales and diary entries will be used to assess panic disorder symptoms and medication side effects. In Phase 3, participants will be randomly assigned to receive either cognitive behavioral therapy (CBT) or sertraline and clonazepam for 12 weeks. All participants will have weekly study visits during Phase 3. Questionnaires and self-report scales will be used to assess participants at the end of Phase 3.

Study hypothesis: Combined selective serotonin reuptake inhibitors (SSRIs) and benzodiazepine treatment, increasing the dose of SSRI, and the addition of cognitive behavioral therapy (CBT) each may have benefits for patients with panic disorder who remain symptomatic after initial treatment with SSRIs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of panic disorder

Exclusion Criteria:

* History of bipolar disorder, schizophrenia, psychosis, or delusional disorders
* Post-traumatic stress disorder diagnosis within 6 months prior to study entry
* Current use of psychotropic medications
* Current use of cognitive behavioral therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1999-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi M. Simon, MD, MSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Simon NM, Otto MW, Worthington JJ, Hoge EA, Thompson EH, Lebeau RT, Moshier SJ, Zalta AK, Pollack MH. Next-step strategies for panic disorder refractory to initial pharmacotherapy: a 3-phase randomized clinical trial. J Clin Psychiatry. 2009 Nov;70(11):1563-70. doi: 10.4088/JCP.08m04485blu. Epub 2009 Oct 6. PMID 19814948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by advertisement and referral to research at the Center for Anxiety and Traumatic Stress Related Disorders at Massachusetts General Hospital.
Pre-assignment Details: 46 participants enrolled, but four participants were lost prior to Phase 1, two due to alcohol abuse and two due to follow-up. Participants were not randomized until the start of Phase 2.
Groups:
- Sertraline / Increased Dose / Medication Optimization: In Phase 1, this group will receive a moderate dose of sertraline (or escitalopram, an equivalent SSRI); In Phase 2, this group will receive an increased dosage of their SSRI; In Phase 3, this group will receive medication optimization, which includes an SSRI and clonazepam
- Sertraline / + Placebo / Cognitive Behavior Therapy Augment.: In Phase 1, this group will receive a moderate dose of sertraline (or escitalopram, an equivalent SSRI); In Phase 2, this group will receive their SSRI plus a placebo; In Phase 3, this group will receive their SSRI plus cognitive behavioral therapy (CBT)
Period: Phase I (Weeks 0 to 6)
Arm/Group | Sertraline / Increased Dose / Medication Optimization | Sertraline / + Placebo / Cognitive Behavior Therapy Augment.
Started | 39 | 0 (In Phase 1, all participants received open label SSRI - no second treatment arm.)
Completed | 21 | 0
Not Completed | 18 | 0
Not completed — Remission | 8 | 0
Not completed — Lost to Follow-up | 6 | 0
Not completed — Loss of Eligibility for Phase 2 | 4 | 0
Period: Phase II (Weeks 6 to 12)
Arm/Group | Sertraline / Increased Dose / Medication Optimization | Sertraline / + Placebo / Cognitive Behavior Therapy Augment.
Started | 11 (Three new participants on Phase 1 endpoint doses of SSRIs entered at Phase 2.) | 13
Completed | 9 | 10
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Remission | 1 | 2
Period: Phase III (Weeks 12 to 24)
Arm/Group | Sertraline / Increased Dose / Medication Optimization | Sertraline / + Placebo / Cognitive Behavior Therapy Augment.
Started | 9 | 10
Completed | 8 | 9
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Change in Panic Disorder Symptoms, Phase 1 (Week 0 - Week 6)
Description: This measure is the change in points between baseline and endpoint scores on the Panic Disorder Severity Scale (PDSS). The PDSS is a 7-item scale with each item rated from 0 (none) to 4 (extreme), for a total score range of 0 to 28 points, and an established interrater reliability of 0.87.
Time Frame: Measured at baseline and after Phase 1 (6 weeks)
Population: Analyses in each study phase were for a modified intent to treat (ITT) sample, defined as all participants who had at least one on-treatment assessment during that phase.
Measure: Mean (Standard Deviation); unit: Points on a scale
Groups:
- Moderate Sertraline Treatment: This group will receive moderate sertraline or escitalopram treatment
Arm/Group | Moderate Sertraline Treatment
Number analyzed (Participants) | 39
Points on a scale | 4.3 (4.3)
Statistical Analysis 1: Comparison: Moderate Sertraline Treatment; Test type: Superiority or Other; p = 0.0000, t-test, 2 sided — Paired t-test between endpoint and baseline PDSS; Degrees of Freedom = 38

2. Primary Outcome: Change in Panic Disorder Symptoms, Phase 2 (Week 6 - Week 12)
Description: as for outcome 1
Time Frame: Measured after Phase 1 (Week 6) and Phase 2 (Week 12)
Measure: Mean (Standard Deviation); unit: Points on a scale
Groups:
- Increased Sertraline: This group will receive an increased dosage of sertraline or escitalopram
- Sertraline Plus Placebo: This group will receive sertraline or escitalopram with a placebo
Arm/Group | Increased Sertraline | Sertraline Plus Placebo
Number analyzed (Participants) | 11 | 13
Points on a scale | 2.36 (3.44) | 2.31 (4.29)
Statistical Analysis 1: Comparison: Increased Sertraline vs Sertraline Plus Placebo; Test type: Superiority or Other; p = 0.97, t-test, 2 sided — T-test of PDSS change score; Degrees of Freedom = 22

3. Primary Outcome: Change in Panic Disorder Symptoms, Phase 3 (Week 12 - Week 24)
Description: as for outcome 1
Time Frame: Measured after Phase 2 (Week 12) and Phase 3 (Week 24)
Measure: Mean (Standard Deviation); unit: Points on a scale
Groups:
- Medication Optimization: This group will receive medication optimization, which includes sertraline or escitalopram with clonazepam
- Augmented Cognitive Behavior Therapy: This group will receive sertraline or escitalopram with cognitive behavioral therapy (CBT)
Arm/Group | Medication Optimization | Augmented Cognitive Behavior Therapy
Number analyzed (Participants) | 9 | 10
Points on a scale | 3.78 (3.80) | 2.9 (3.63)
Statistical Analysis 1: Comparison: Medication Optimization vs Augmented Cognitive Behavior Therapy; Test type: Superiority or Other; p = 0.061, t-test, 2 sided — T-test of PDSS change between baseline and endpoint of Phase 3; Degrees of Freedom = 17

ADVERSE EVENTS:
Groups:
- Phase I: Sertraline: In Phase 1, this group will receive a moderate dose of sertraline (or escitalopram, an equivalent SSRI).
Arm/Group | Phase I: Sertraline | Phase II: Cont. SSRI Plus Placebo OR Increased Dose SSRI Alone | Phase III: Cont. Medication Plus CBT OR SSRI and Clonazepam
Serious Adverse Events (participants affected / at risk) | 2/39 | 0/24 | 3/19
Other Adverse Events (participants affected / at risk) | 33/39 | 21/24 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Sertraline (N=39) | Phase II: Cont. SSRI Plus Placebo OR Increased Dose SSRI Alone (N=24) | Phase III: Cont. Medication Plus CBT OR SSRI and Clonazepam (N=19)
Patient admitted to inpatient rehabiliation center for alcohol abuse (General disorders) | 0 (0) | 0 (0) | 2 (2) — 1. A patient receiving Sertraline and Clonazepam was admitted to rehab center for alcohol abuse. 2. A patient who completed Phase III of the study, receiving Sertraline and Clonazepam, was admitted to rehab center for alcohol abuse.
Patient admitted to the hospital after experiencing symptoms similar to panic attacks. (General disorders) | 1 (1) | 0 (0) | 0 (0) — This patient in Phase I of the study was admitted to the hospital after experiencing symptoms similar to, but more intense than panic attacks. The subject had not yet initiated study medication when the event occurred.
Patient was in a motorcycle accident of unknown etiology (General disorders) | 0 (0) | 0 (0) | 1 (1) — This patient completed Phase III of the study (Sertraline and Clonazepam), and was involved in a motorcycle accident months after study completion. There is no evidence to indicate that the medication was related to the accident.
Patient was found to have blockage of one cardiac vessel (General disorders) | 1 (1) | 0 (0) | 0 (0) — Patient presented to the emergency room with sudden onset leg pain and was found to have blockage of one cardiac vessel. These symptoms were determined to be unrelated to the study medication (escitalopram); thus, her study treatment was not altered.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Sertraline (N=39) | Phase II: Cont. SSRI Plus Placebo OR Increased Dose SSRI Alone (N=24) | Phase III: Cont. Medication Plus CBT OR SSRI and Clonazepam (N=19)
Gastrointestinal distress (Gastrointestinal disorders) | 19 (19) | 7 (7) | 6 (6)
Headache (General disorders) | 16 (16) | 7 (7) | 6 (6)
Nausea or Vomiting (General disorders) | 15 (15) | 0 (0) | 0 (0)
Jitteriness or Restlesness (General disorders) | 12 (12) | 4 (4) | 0 (0)
Insomnia (General disorders) | 11 (11) | 4 (4) | 0 (0)
Sedation (General disorders) | 0 (0) | 6 (6) | 4 (4)
Dizziness (General disorders) | 0 (0) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Power in Phase 2 limited detection to a large effect size. High drop-out for increased SSRI dose may indicate poor tolerability. Effectiveness of adding an SSRI to initial CBT was unexamined, limiting generalization to community treatment decisions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No